CLINICAL TRIAL: NCT05334472
Title: Real World Study to Evaluate Patient and Care Partner Ratings on Early Experience of Injection and Device for KESIMPTA® (Ofatumumab) Indicated for Multiple Sclerosis
Brief Title: A Survey to Evaluate Early Experience From Patient and Care Partner on Injection and Device for KESIMPTA® Indicated for Multiple Sclerosis
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: COMB157GUS13
Record Dates: First submitted 2022-03-21; First posted 2022-04-19 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; MS; NIS; KESIMPTA; ofatumumab
MeSH Terms: conditions — Multiple Sclerosis | interventions — ofatumumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Kesimpta: Patients or caregivers of patients administered Kesimpta
  Interventions: Other: Kesimpta

INTERVENTIONS:
Other: Kesimpta — There was no treatment allocation. Patients administered Kesimpta by prescription that started before inclusion of the patient into the study were enrolled.
  Other Names: ofatumumab

SUMMARY:
This was a US-based, observational cross-sectional study with primary data collection via questionnaires directly administered to patients with MS receiving KESIMPTA and care partners of patients with MS (formal or informal)receiving KESIMPTA.

DETAILED DESCRIPTION:
The study aimed to enroll ninety-four (94) patients/care partners. The time period for enrollment was dependent on the uptake of KESIMPTA in the real-world.

Data collected for the study was obtained directly from the patient/care partner within the web-based database: De-identified data was stored on a secure server and transferred for analysis. Responses from the patient and care partner surveys were pooled for analysis of study endpoints.

ELIGIBILITY:
Patients with MS Inclusion Criteria:

* Adult aged eighteen (18) years of age or over at the time of the survey
* Prescribed KESIMPTA within the prior 12 months and currently self-administering treatment using the Sensoready® pen
* MS diagnosis based on 2017 McDonald criteria

Care Partner Inclusion Criteria:

* Adult aged eighteen (18) years of age or over
* Formal or informal care partner of patient with MS prescribed KESIMPTA within the prior 12 months
* Is currently administering KESIMPTA using the Sensoready® pen on their patient's behalf

Patients with MS Exclusion Criteria:

* Previously used injection as a part of inclusion in any ofatumumab (OMB) randomized clinical trial
* Active Hepatitis B virus (HBV)
* Cognitive impairment that would impact their ability to participate in a survey study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: To ensure a representative sample of patients with MS, the patient study population will include patients who are new to the use of injectable treatments for MS, as well as those with use of other injectable MS treatments prior to initiation of KESIMPTA using the Sensoready® pen.
  Patients care partner (formal or informal) may also be eligible for study participation.
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2021-11-24 (Actual); Primary Completion 2023-02-15 (Actual); Study Completion 2023-02-15 (Actual)

PRIMARY OUTCOMES:
Proportion of respondents in top two rating categories for device satisfaction on use of KESIMPTA Sensoready | Up to 6 months, at the time of survey completion
  Proportion of respondents (patients and care partners) in top two rating categories (satisfied and extremely satisfied) for device satisfaction on use of KESIMPTA Sensoready®

SECONDARY OUTCOMES:
Proportion of patients by US region of residence | Up to 6 months, at the time of survey completion
  Census US geographic region of residence (Northeast, Midwest, South, or West)
Proportion of patients by educational level | Up to 6 months, at the time of survey completion
  Proportion of patients by educational level was collected
Patients Determined Disease Steps (PDDS) | Up to 6 months, at the time of survey completion
  PDDS was used as a proxy to Expanded Disability Status Scale (EDSS). People were asked to choose one out of nine options that best describes how well they walk. 0 is "normal" and 8 is "bedridden."
General Health | Up to 6 months, at the time of survey completion
  Participants were asked "How is your general health today?" and they had to choose one out of five options that best describes how well they feel from "Poor", "Fair" ,"Good", "Very Good" to "Excellent".
Proportion of patients by Multiple Sclerosis Phenotype | Up to 6 months, at the time of survey completion
  Proportion of patients by Multiple Sclerosis Phenotype was collected:
  * RRMS: Relapsing-Remitting Multiple Sclerosis
  * SPMS: Secondary Progressive Multiple Sclerosis
Proportion of patients with co-morbidities | Up to 6 months, at the time of survey completion
  Proportion of patients with co-morbidities was collected
Importance of healthcare provider (HCP) instructions for first injection | Up to 6 months, at the time of survey completion
  Participants were asked to rate their level of agreement with each statement related to their first Kesimpta injection. 1) I felt it was essential to have a healthcare provider instruct me on how to perform my first KESIMPTA injection using the Sensoready® pen, 2) I felt I needed to have a healthcare provider watch me administer my first KESIMPTA injection using the Sensoready® pen, and 3) I felt comfortable receiving instructions from my healthcare provider in the clinic on how to administer my first KESIMPTA injection using the Sensoready® pen and did not need my healthcare provider to be present to administer it at home.
  Participants were asked to choose five options toward each statement from "Strongly Disagree" to "Strongly Agree".
Level of anxiety with injections, in general | Up to 6 months, at the time of survey completion
  Participants were asked "Using a scale of 0 to 10, 0 being Not at All Confident and 10 being Extremely Confident, how confident do you feel about your ability to administer KESIMPTA using the Sensoready® pen on your own?"
Proportion of patients performing preparation activities for injection | Up to 6 months, at the time of survey completion
  Proportion of patients performing preparation activities for injection:
  * Time to take KESIMPTA Sensoready® pen out of the refrigerator and allow it to reach room temperature prior to injection (minutes) (step A)
  * Time to perform the injection including picking up the Sensoready® pen, injecting and disposing in the sharps container (minutes) (step B)
Proportion of participants by site of administration | Up to 6 months, at the time of survey completion
  Proportion of participants by site of administration was collected:
  * thigh
  * abdomen
  * upper outer arm
Proportion of participants by individual medication as previous Disease Modifying Therapy (DMT) | Up to 6 months, at the time of survey completion
  Proportion of participants by individual medication as previous Disease Modifying Therapy (DMT) was collected among DMT experienced patients
Proportion of patients who are DMT naïve or experienced | Up to 6 months, at the time of survey completion
  Proportion pf patients who are DMT naïve or experienced was collected.
Proportion of participants by reasons for starting KESIMPTA | Up to 6 months, at the time of survey completion
  Proportion of participants by reasons for starting KESIMPTA was collected:
  * ease of dosing schedule
  * avoidance of infusion clinics
  * at home convenience
  * enhanced efficacy and safety profile
  * HCP recommendation
  * lack of insurance coverage for other DMTs
  * Other
Proportion of participants by reasons to switch from most recent therapy | Up to 6 months, at the time of survey completion
  Proportion of participants by reasons to switch from most recent therapy (insurance, lack of efficacy/wear off effect, side-effects and tolerability, adherence concerns etc.) was collected among DMT experienced patients.
Proportion of patients agreeing with the attributes of the device Usability Characteristics during self-administration | Up to 6 months, at the time of survey completion
  Percentage of patients who agree with each attribute of the device Usability Characteristics during self-administration, based on patient self-report was collected:
  * Overall ease of use
  * Device ergonomics ("feeling" in the hand )
  * Steps for preparing and using device
  * Time required for preparation and use of device
  * Convenience/Flexibility for travel with device
Patient Confidence | Up to 6 months, at the time of survey completion
  Percentage o patients who agree with each attribute regarding confidence, based on patient self-report, was collected:
  * Confidence to self-administer KESIMPTA using the device
  * Intention to continue use of device
  * Recommendation of KESIMPTA device use to others
  * Ease of KESIMPTA's monthly dosing schedule
Overall device satisfaction by treatment duration | Up to 6 months, at the time of survey completion
  Overall device satisfaction. Participants choose between five options from 1: Extremely Dissatisfied, 2 Dissatisfied, 3: Neither Satisfied nor Dissatisfied, 4: Satisfied, 5: Extremely Satisfied. The higher score means a better overall devise satisfaction.
Overall device satisfaction score of the study participants by DMT experience | Up to 6 months, at the time of survey completion
  Percentage of patients by overall satisfaction score (extremely dissatisfied, dissatisfied, neither satisfied nor dissatisfied, satisfied, extremely satisfied) by DMT experience

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, East Hanover, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Results for COMB157GUS13 that is getting linked from the Novartis Clinical Trials Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=18144